CLINICAL TRIAL: NCT04729855
Title: Association of Autophagy-related Genes ,LncRNA and SNPs With Colorectal Cancer in Egyptian Population
Status: Completed | Type: Observational
Sponsor: Esraa Hassan,MD (Other)
Collaborators: South Egypt Cancer Institute (Other)
Responsible Party: Sponsor-Investigator, Esraa Hassan,MD, Principle investigator, Assiut University
Organization: Assiut University (Other)
Other Study IDs: Esraa Hassan MD Protocol
Record Dates: First submitted 2021-01-24; First posted 2021-01-29 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Colo-rectal Cancer
Keywords: Colorectal cancer, HOTTIP
MeSH Terms: conditions — Colonic Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — EDTA (ethylene diamine tetra acetic acid)coated fresh blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- colorectal cancer patients: Colorectal cancer patients( n = 30 ) from stage I-III with the following criteria:-
  a. Inclusion criteria:
  * No sex predilection.
  * Age (25-65 yr).
  * Colorectal carcinoma confirmed by histopathological examination
  Interventions: Diagnostic Test: PBMCs and Tissue expression of HOTTIP ,EIF4EBP1 and serum SNP HOTTIP rs1859168
- Healthy controls ( n = 30): matched as regarding age and sex as much as possible with cases.
  Interventions: Diagnostic Test: PBMCs and Tissue expression of HOTTIP ,EIF4EBP1 and serum SNP HOTTIP rs1859168

INTERVENTIONS:
Diagnostic Test: PBMCs and Tissue expression of HOTTIP ,EIF4EBP1 and serum SNP HOTTIP rs1859168 — 5 ml fresh blood sample, normal and CRC tissue

SUMMARY:
1. Determination of expression level of HOTTIP and EIF4EBP1(Eukaryotic translation initiation factor 4E-binding protein 1) .
2. Investigation of the SNP HOTTIP rs1859168 and it's association with CRC susceptibility.
3. Correlation of the expression of these genes with various stages of CRC to determine the prognostic value of each of them.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is a common digestive tract tumor 1.It is the third leading cause of death in the world. Overall 5-year survival rate is less than 40%, and the occurrence is rising 2. However, the prognosis and therapy have not been significantly improved. Therefore, a proper selection of patients for aggressive treatment is necessary, new therapeutic and prognostic strategies are urgently needed 3.

Autophagy is a pathway for self-digestion, in which unwanted cytoplasmic components are recycled 4.In normal conditions, autophagy is essential for cellular homeostasis 5. Autophagy has dual roles in cancer cells, stimulation or suppression , with effects on progression and oncogenesis 6.Recent research established that autophagy is important target for controlling cancer depending on stage and type of tumor 7.Diverse molecular mechanisms contribute to cancer cells resistance to treatment 8.Among these mechanisms , autophagy appears to be critical 9.

EIF4EBP1 (Eukaryotic translation initiation factor 4E-binding protein 1) is encoded by EIF4EBP1 gene.It acts as an effector in mTOR (mammilian target of rapamycin) pathway which on activation ,EIF4EBP1 is phosphorylated promoting cell proliferation 10. Studies have suggested that EIF4EBP1 promotes carcinogenesis as in hepatocellular carcinoma .However, its role in CRC have not been elucidated 10.

Long non-coding RNAs (lncRNAs) are group of RNA , 200 nucleotides in length 11,. Expression of lncRNAs has been discovered in multiple tumors, acting as oncogenes. 'HOXA(hydrogenase transcriptional regulatory protein) transcript at the distal tip' (HOTTIP) has received attention lately.It is up-regulated in CRC tissue, regulating genes via epigenetic modification. Therefore, it might be a candidate for cancerization and therapy of CRC 12.

Expression of lncRNAs could be affected by single nucleotide polymorphisms (SNPs), the most common genetic variation in human genomes13. rs1859168 was reported as a potential functional polymorphism on HOTTIP that alters its expression level 14.. Also, it was recently reported that HOTTIP enhances interleukin 6 expression, which potentiates immune escape of cancer cells 15.

ELIGIBILITY:
Inclusion Criteria:

* No sex predilection.
* Age (25-65 yr).
* Colorectal carcinoma confirmed by histopathological examination

Exclusion Criteria:

* -patients who received any treatment.
* Cases with other organ cancers.
* History of chemotherapy and radiotherapy.
* Systemic diseases such as renal failure, diabetes mellitus, and hypertension.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Healthy controls ( n = 30) matched as regarding age and sex as much as possible with cases.
  -Colorectal cancer patients( n = 30 ) from stage I-III with the following criteria:-
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2022-04-15 (Actual); Primary Completion 2023-05-20 (Actual); Study Completion 2024-09-20 (Actual)

PRIMARY OUTCOMES:
HOTTIP gene expression | 2 years
  Estimation of expression level of HOTTIP in peripheral blood mononuclear cells and tissue aiming to use as possible less invasive prognostic markers for colorectal cancer.

SECONDARY OUTCOMES:
EIF4EBP | 2 years
  Estimation of expression level of EIF4EBP in peripheral blood mononuclear cells and tissue

CONTACTS AND LOCATIONS:
Overall Officials: Esraa H Mohamed, Master, Principal Investigator — Assistant lecturer of Medical Microbiology and Immunology
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
all researchers will have access to individual patient data with preserving confidentiality

REFERENCES:
- [Background] Chisanga D, Keerthikumar S, Pathan M, Ariyaratne D, Kalra H, Boukouris S, Mathew NA, Al Saffar H, Gangoda L, Ang CS, Sieber OM, Mariadason JM, Dasgupta R, Chilamkurti N, Mathivanan S. Colorectal cancer atlas: An integrative resource for genomic and proteomic annotations from colorectal cancer cell lines and tissues. Nucleic Acids Res. 2016 Jan 4;44(D1):D969-74. doi: 10.1093/nar/gkv1097. Epub 2015 Oct 22. PMID 26496946
- [Background] Vorobiova OA. [Participation of the supraoptic nucleus of the anterior hypothalamus in controlling the gonadotropic functions of the pituitary]. Fiziol Zh. 1974 May-Jun;20(3):334-8. No abstract available. Ukrainian. PMID 4466671
- [Background] Katheder NS, Khezri R, O'Farrell F, Schultz SW, Jain A, Rahman MM, Schink KO, Theodossiou TA, Johansen T, Juhasz G, Bilder D, Brech A, Stenmark H, Rusten TE. Microenvironmental autophagy promotes tumour growth. Nature. 2017 Jan 19;541(7637):417-420. doi: 10.1038/nature20815. Epub 2017 Jan 11. PMID 28077876
- [Background] Rahman MA, Rhim H. Therapeutic implication of autophagy in neurodegenerative diseases. BMB Rep. 2017 Jul;50(7):345-354. doi: 10.5483/bmbrep.2017.50.7.069. PMID 28454606
- [Background] Uddin MS, Stachowiak A, Mamun AA, Tzvetkov NT, Takeda S, Atanasov AG, Bergantin LB, Abdel-Daim MM, Stankiewicz AM. Autophagy and Alzheimer's Disease: From Molecular Mechanisms to Therapeutic Implications. Front Aging Neurosci. 2018 Jan 30;10:04. doi: 10.3389/fnagi.2018.00004. eCollection 2018. PMID 29441009
- [Background] Avalos Y, Canales J, Bravo-Sagua R, Criollo A, Lavandero S, Quest AF. Tumor suppression and promotion by autophagy. Biomed Res Int. 2014;2014:603980. doi: 10.1155/2014/603980. Epub 2014 Sep 18. PMID 25328887
- [Background] Abdullah LN, Chow EK. Mechanisms of chemoresistance in cancer stem cells. Clin Transl Med. 2013 Jan 17;2(1):3. doi: 10.1186/2001-1326-2-3. PMID 23369605
- [Background] Ojha R, Bhattacharyya S, Singh SK. Autophagy in Cancer Stem Cells: A Potential Link Between Chemoresistance, Recurrence, and Metastasis. Biores Open Access. 2015 Jan 1;4(1):97-108. doi: 10.1089/biores.2014.0035. eCollection 2015. PMID 26309786
- [Background] Cha YL, Li PD, Yuan LJ, Zhang MY, Zhang YJ, Rao HL, Zhang HZ, Zheng XF, Wang HY. EIF4EBP1 overexpression is associated with poor survival and disease progression in patients with hepatocellular carcinoma. PLoS One. 2015 Feb 6;10(2):e0117493. doi: 10.1371/journal.pone.0117493. eCollection 2015. PMID 25658620
- [Background] Bonasio R, Shiekhattar R. Regulation of transcription by long noncoding RNAs. Annu Rev Genet. 2014;48:433-55. doi: 10.1146/annurev-genet-120213-092323. Epub 2014 Sep 18. PMID 25251851
- [Background] Wang KC, Yang YW, Liu B, Sanyal A, Corces-Zimmerman R, Chen Y, Lajoie BR, Protacio A, Flynn RA, Gupta RA, Wysocka J, Lei M, Dekker J, Helms JA, Chang HY. A long noncoding RNA maintains active chromatin to coordinate homeotic gene expression. Nature. 2011 Apr 7;472(7341):120-4. doi: 10.1038/nature09819. Epub 2011 Mar 20. PMID 21423168
- [Background] Lv Z, Xu Q, Yuan Y. A systematic review and meta-analysis of the association between long non-coding RNA polymorphisms and cancer risk. Mutat Res Rev Mutat Res. 2017 Jan-Mar;771:1-14. doi: 10.1016/j.mrrev.2016.10.002. Epub 2016 Nov 5. PMID 28342449
- [Background] Hu P, Qiao O, Wang J, Li J, Jin H, Li Z, Jin Y. rs1859168 A > C polymorphism regulates HOTTIP expression and reduces risk of pancreatic cancer in a Chinese population. World J Surg Oncol. 2017 Aug 17;15(1):155. doi: 10.1186/s12957-017-1218-0. PMID 28818070
- [Background] Shang A, Wang W, Gu C, Chen C, Zeng B, Yang Y, Ji P, Sun J, Wu J, Lu W, Sun Z, Li D. Correction to: Long non-coding RNA HOTTIP enhances IL-6 expression to potentiate immune escape of ovarian cancer cells by upregulating the expression of PD-L1 in neutrophils. J Exp Clin Cancer Res. 2020 Dec 4;39(1):272. doi: 10.1186/s13046-020-01755-z. PMID 33272287